CLINICAL TRIAL: NCT03096561
Title: A Comparative Study of Serum Potassium Rate Between Peripheral and Central Venous Sample Collection in Patients With Hypothermia Related Cardiac Arrest
Brief Title: Measurement of Serum Potassium Rate During Accidental Hypothermia.
Acronym: Kai+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other); Centre Hospitalier Universitaire Vaudois (Other); Emergency Department, Hospital of Valais, Sion (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N° ID-RCB: 2016-A01762-49
Record Dates: First submitted 2017-03-16; First posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Accidental Hypothermia; Hyperkalemia; Cardiac Arrest
MeSH Terms: conditions — Hypothermia; Hyperkalemia; Heart Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypothermia related cardiac arrest (Other): blood draw from three different vessels punctured in the emergency room (central vein, peripheral vein, artery) and comparison of potassium rate and other biological values between the different sites of blood draw and two different measuring techniques (laboratory vs. blood gas analyser)
  Interventions: Diagnostic Test: blood draw from three different vessels

INTERVENTIONS:
Diagnostic Test: blood draw from three different vessels — Patient in cardiac-arrest and cold exposure, diagnostic test: blood draw from three different vessels (central vein, artery, peripheral vein) and measuring of PR

SUMMARY:
Serum Potassium Rate (PR) is a key indicator for medical management of patients with accidental hypothermia particularly for hypothermia related cardiac arrest (CA).

Experts recommend a cut-off value for PR of 12 mmol/l for all hypothermic victims and 8 mmol/l for avalanche casualties. Any patient presenting a PR lower than the cut-off value should be considered for Extracorporeal Rewarming. This therapeutic strategy is vital for patient survival.

However, there is no consensus about what type of vessels should be punctured in order to obtain an accurate potassium rate and what type of measurement technics should be used to measure this potassium rate.

The investigators hypothesize that potassium rate in these patients will differ by 1 mmol/l in blood samples collected from a peripheral vein in contrast to a central vein.

The investigators study is a prospective observational, multicentre study.

ELIGIBILITY:
Inclusion Criteria:

* Hypothermia related cardiac arrest
* Age > 18 years
* Core temperature < 30° C measured in oesophagus at hospital admission

Exclusion Criteria:

* Age < 18 years
* Known condition of pregnancy or breastfeeding women
* Evidence of trauma-related cardiac arrest
* Cardiac arrest in which reanimation is not justified (frozen body, final stadium of an incurable disease, advance health care directive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-11-14 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of potassium rate in central venous blood and blood from a peripheral vein (measured in mmol/l) | 24 hours
  Comparison of PR in central venous blood and blood from a peripheral vein (measured in mmol/l)

SECONDARY OUTCOMES:
Comparison of potassium rate in venous and arterial blood (measured in mmol/l) | 24 hours
  Comparison of potassium rate in venous and arterial blood (measured in mmol/l)
Comparison of potassium rate from laboratory analysis and at bedside via blood gas analyser (measured in mmol/l) | 24 hours
  Comparison of potassium rate from laboratory analysis and at bedside via blood gas analyser (measured in mmol/l)
Comparison of the time difference between laboratory analysis and blood gas analyzer at bed side (measured in minutes) | 24 hours
  Comparison of the time difference between laboratory analysis and blood gas analyzer at bed side (measured in minutes)
Survival and neurological outcome as measured by the Cerebral Performance Category Scale | 3 months
  Survival and neurological outcome as measured by the Cerebral Performance Category Scale
Study of biological parameters to calculate the Strong Ion Gap (measured in mEq/l) according to the Stewart Approach | 24 hours
  1. For each sample, the apparent strong ion difference (SIDa) will be calculated as SIDa =(Na+ +K+ +Ca2+ +Mg2+)-(Cl- +Lac-)
  2. The amount of weak plasma acid (A-) will be calculated as:
     A- = [Alb] × (0.123 × pH - 0.631) + [PO4] × (0.309 × pH - 0.469)
  3. The effective strong ion difference (SIDe) will be calculated as:
  SIDe = 1000 × 2.46 × 10-11 × PaCO2/(10-pH) + [A-]
  To quantify unmeasured charges, the SIG will be calculated as:
  SIG = SIDa - SIDe

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital Vaudois, Lausanne, Valais
  - Hospital of Valais, Sion, Valais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pasquier M, Blancher M, Buse S, Boussat B, Debaty G, Kirsch M, de Riedmatten M, Schoettker P, Annecke T, Bouzat P. Intra-patient potassium variability after hypothermic cardiac arrest: a multicentre, prospective study. Scand J Trauma Resusc Emerg Med. 2019 Dec 16;27(1):113. doi: 10.1186/s13049-019-0694-3. PMID 31842931